CLINICAL TRIAL: NCT06455098
Title: Assessment of Safety and Effectiveness in Treatment Management of Paroxysmal Atrial Fibrillation With the BWI Pulsed Field Ablation System With OMNYPULSE™ Catheter
Brief Title: A Study of Assessment on Safety and Effectiveness of BWI Pulsed Field Ablation With OMNYPULSE Catheter for the Treatment of Paroxysmal Atrial Fibrillation (PAF)
Acronym: OMNY-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI202303; BWI202303 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Pulsed Field (PF) Ablation System (Experimental): Participants with PAF will undergo pulsed field ablation procedure with the OMNYPULSE™ catheter in combination with TRUPULSE™ generator for PVI and to deliver pulsed field (PF) energy for treatment of atrial fibrillation. Study participants will be followed for 12 months after the study index procedure.
  Interventions: Device: OMNYPULSE™ Catheter with the TRUPULSE Generator

INTERVENTIONS:
Device: OMNYPULSE™ Catheter with the TRUPULSE Generator — OMNYPULSE™ Catheter and TRUPULSE™ Generator will be used for PF ablation.

SUMMARY:
The purpose of this study is to demonstrate the safety and 12-month effectiveness of the BWI OMNYPULSE™ pulsed field ablation (PFA) platform for pulmonary vein isolation (PVI) in the treatment of participants with symptomatic paroxysmal atrial fibrillation (PAF), an irregular heart rate that causes abnormal blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic paroxysmal AF with:

  1. At least two symptomatic AF episodes within last six months from enrollment
  2. At least one electrocardiographically documented AF episode within twelve months prior to enrollment
* Failed at least one Class I or Class III antiarrhythmic drug
* Willing and capable to provide consent
* Able and willing to comply with all pre-, post- and follow-up testing and requirements

Exclusion Criteria:

* Previously diagnosed with persistent AF (greater than [>] 7 days in duration)
* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
* Previous surgical or catheter ablation for AF
* Patients known to require ablation outside the PV ostia and outside the CTI region.
* Documented severe dilatation of the left atrium (LAD>50 mm) antero-posterior diameter on imaging within 6 months prior to enrollment
* Documented left atrium (LA) thrombus by imaging within 48 hours of the procedure
* Documented severely compromised left ventricular ejection fraction (LVEF <40%) by imaging within 6 months prior to enrollment
* Uncontrolled heart failure or New York Heart Association (NYHA) Class III or IV
* History of blood clotting, bleeding abnormalities or contraindication to anticoagulation (heparin, warfarin, or dabigatran)
* Documented thromboembolic event (including transient ischemic attack or TIA) within the past 6 months
* Previous Percutaneous Coronary Intervention (PCI)/ myocardial infarction [MI] within the past 2 months
* Coronary Artery Bypass Grafting (CABG) surgery within the past 6 months
* Valvular cardiac surgical/percutaneous procedure
* Unstable angina within 6 months
* Anticipated cardiac transplantation, cardiac surgery, or other major surgery within the next 12 months
* Significant pulmonary disease or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
* Prior diagnosis of pulmonary vein stenosis
* Pre-existing hemi diaphragmatic paralysis
* Acute illness, active systemic infection, or sepsis
* Presence of intracardiac thrombus, myxoma, tumor, interatrial baffle or patch or other abnormality that precludes catheter introduction or manipulation
* Severe mitral regurgitation
* Presence of an implanted pacemaker or Implantable Cardioverter-Defibrillator (ICD) or other implanted metal cardiac device (other than coronary stents) that may interfere with the PF energy field)
* Presence of a condition that precludes vascular access
* Current enrollment in an investigational study evaluating another device or drug
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal), lactating, or who are of child-bearing age and plan on becoming pregnant during the course of the clinical investigation
* Life expectancy less than 12 months
* Presenting contra-indications for the devices used in the study, as indicated in the respective Instructions for Use (IFU)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Primary Adverse Events (PAEs) | 7 days post-procedure
  Number of participants with PAEs (within 7 days following the ablation procedure unless otherwise indicated) will be reported. PAEs will include the following adverse events: esophageal perforating complications (atrio-esophageal fistula, esophago-pericardial fistula), phrenic nerve paralysis (permanent), cardiac tamponade/perforation, pulmonary vein stenosis (PVS), device or procedure related death, stroke/cerebrovascular accident (CVA), major vascular access complication/bleeding, thromboembolism, myocardial infarction, transient ischemic attack (TIA), pericarditis, heart block, pulmonary edema (respiratory insufficiency) and vagal nerve injury/gastroparesis.
Number of Participants Reporting Freedom from Documented (Symptomatic and Asymptomatic) Atrial Tachyarrhythmia (Atrial Fibrillation [AF], Atrial Tachycardia [AT] or Atrial Flutter [AFL] of Unknown Origin) Episodes | Day 91 to Day 365 post-procedure
  Number of participants reporting freedom from documented (symptomatic and asymptomatic) atrial tachyarrhythmia (AF, AT, or AFL of unknown origin) episodes of >= 30 seconds based on sponsor provided transtelephonic monitoring (TTM) or holter device or continuous on standard 12-lead electrocardiogram (ECG) data during the effectiveness evaluation period will be reported.

SECONDARY OUTCOMES:
Change from Baseline in Atrial Fibrillation Effect on Quality of Life (AFEQT) Total Score | Baseline, Month 12
  The AFEQT uses a questionnaire to evaluate symptoms, daily activities and treatment concerns participants have related to atrial fibrillation. An overall AFEQT score ranges from 0 to 100. A score of 0 corresponds to complete disability (or responding "extremely" difficult to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered). A positive change in score corresponds to improvement in AF symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster, Inc. Clinical Trial, Study Director — Biosense Webster, Inc.
Locations (46):
- United States (43):
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Mills Peninsula Health Services, Burlingame, California
  - Scripps Clinic/Prebys Cardiovascular Institute, La Jolla, California
  - Cardiovascular Associates of Marin, Larkspur, California
  - Loma Linda Medical Center, Loma Linda, California
  - Hoag Memorial Hospital, Newport Beach, California
  - San Diego Cardiac Center, San Diego, California
  - California Pacific Medical Center- Sutter Health, San Francisco, California
  - Providence Saint John s Health Center, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Ascension St. Vincent's, Jacksonville, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - HCA Florida Mercy Hospital, Miami, Florida
  - NCH Healthcare, Naples, Florida
  - Advent Health Orlando, Orlando, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - NorthShore University Medical Center, Glenview, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General, Boston, Massachusetts
  - Brigham And Women's Hospital, Boston, Massachusetts
  - Beaumont Health Systems, Royal Oak, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - New York Presbyterian - Weill Cornell Medical Ctr, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - WakeMed Heart & Vascular, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Texas Heart Institute, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Fairfax Medical Campus- Inova Heart and Vascular Institute, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Canberra Heart Rhythm, Garran
  - Royal Melbourne Hospital, Parkville

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency